CLINICAL TRIAL: NCT02523092
Title: Use of CXCL9 as a Biomarker of Acthar Efficacy
Acronym: Acthar
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-17300
Record Dates: First submitted 2015-08-10; First posted 2015-08-14 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Sarcoidosis
Keywords: sarcoidosis; Acthar; CXCL9; chemokine ligand 9
MeSH Terms: conditions — Sarcoidosis | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acthar gel (Experimental): After a 4-week period of baseline monitoring, Acthar gel will be administered by intramuscular or subcutaneous injection. Initial dosing will be 40 U every 72 hours (or twice per week) for 4 weeks. Dosage will then be increased to 80 U with similar frequency for 8 weeks and up to 16 weeks.
  Interventions: Drug: Acthar gel

INTERVENTIONS:
Drug: Acthar gel — Acthar gel given IM or SQ as per package insert
  Other Names: Acthar

SUMMARY:
The objective is this study is to test whether use of Acthar gel in the context of sarcoidosis will lead to improved symptoms and lung function and correlate with decreased levels of predictive blood biomarkers, like chemokine ligand 9 (CXCL9).

DETAILED DESCRIPTION:
The investigators will test whether Acthar gel's anti-inflammatory properties will modulate immune cells and lead to decreases in blood biomarkers and improvements in clinical parameters. Specific Aim 1 will examine the levels of the predictive biomarker, chemokine ligand 9 (CXCL9), and related transcripts, and determine whether they decrease in participants over time while taking Acthar. Specific Aim 2 will test whether the biologic changes measured in blood correlate to clinical markers, including lung function and symptom scores. Since the investigators have found that CXCL9 predicts clinical course, they hypothesize that CXCL9 transcript levels in the blood will decrease over time in pulmonary sarcoidosis participants whose clinical outcome measures improve with Acthar.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven diagnosis of sarcoidosis with demonstrated pulmonary involvement
* Refractoriness to or intolerance of immunosuppressive agents like prednisone or methotrexate

Exclusion Criteria:

* Smoking
* Cancer
* Chronic infections (e.g. tuberculosis, viral, fungal, bacterial)
* Inflammatory conditions
* Coexisting lung disease
* Congestive heart failure
* Uncontrolled hypertension
* Recent surgery
* Active peptic ulcers
* Osteoporosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Decrease in blood CXCL9 levels by 50% | within 6 months

SECONDARY OUTCOMES:
Improvement in FVC by 5% of predicted | within 6 months
Improvement in dyspnea score | within 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Laura Koth, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Su R, Li MM, Bhakta NR, Solberg OD, Darnell EP, Ramstein J, Garudadri S, Ho M, Woodruff PG, Koth LL. Longitudinal analysis of sarcoidosis blood transcriptomic signatures and disease outcomes. Eur Respir J. 2014 Oct;44(4):985-93. doi: 10.1183/09031936.00039714. Epub 2014 Aug 19. PMID 25142485
- See also: Homepage for the Sarcoidosis Research Program at the University of California, San Francisco — http://sarcoidosis.ucsf.edu/